CLINICAL TRIAL: NCT00910312
Title: Evaluation of Safety and Feasibility of the ICE-SENSE™, a Cryotherapy Device for Office-based Ultrasound-guided Treatment of Breast Fibroadenoma
Brief Title: ICE-SENSE™ Cryotherapy for Breast Fibroadenoma Trial
Acronym: ICE-CRYSTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IceCure Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-03; version 5.0
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2016-04

CONDITIONS: Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast Fibroadenoma (Experimental)
  Interventions: Device: Ice-Sense

INTERVENTIONS:
Device: Ice-Sense — Ice-Sense Cryoprobe

SUMMARY:
The purpose of this study is to determine whether the Ice-Sense, a novel cryotherapy system (a system that freezes tissues), is safe and effective in the treatment of benign breast tumors such as fibroadenoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient is above 18 years old.
* Patient has breast fibroadenoma, proven by biopsy (Core Biopsy).
* Patient's fibroadenoma can be visualized with ultrasound.
* Patient's fibroadenoma size is between 0.5cm and 3cm at its largest dimension.
* Patient is able to visit the clinic as needed during the 12-month follow-up period following the cryoablation procedure.
* The patient has been informed of the study and agrees to its provisions, and has signed an IRB/EC approved written informed consent, including data privacy authorization.

Exclusion Criteria:

* Patients with history of breast cancer.
* Women with known pregnancy.
* Patients with superficial fibroadenoma very close to the skin.
* Patient has undergone major surgery within the previous 12 weeks.
* Patients with any terminal illness, or with a life expectancy <2 year.
* Patients carrying contagious diseases such as Tuberculosis Hepatitis or AIDS.
* Patient participating in other trials using drugs or devices.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
engulfment of the tumor by the ice-ball as seen under ultrasound imaging | during the procedure

SECONDARY OUTCOMES:
any device related adverse events or complications that may occur | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Klein, Dr., Principal Investigator
Locations (4):
- Oncogynecological Center, Department of Obstetrics and Gynecology, First Faculty of Medicine, Charles University in Prague and General University Hospital in Prague, Prague, Czechia
- Germany (2):
  - Department of Obstetrics and Gynecology, University Hospital of Heidelberg, Heidelberg
  - Department of Obstetrics and Gynecology, University Hospital of Tuebingen, Tübingen
- Assuta medical centers, Haifa, Israel